CLINICAL TRIAL: NCT00627835
Title: A Phase I Dose Escalation Trial of Neoadjuvant Sorafenib and Concurrent Sorafenib, Cisplatin and Radiation in Locally Advanced Squamous Cell Carcinomas of the Head and Neck (SCCHN)
Brief Title: Dose Escalation Trial of Neoadjuvant Sorafenib and Concurrent Sorafenib, Cisplatin and Radiation in Locally Advanced Squamous Cell Carcinomas of the Head and Neck (SCCHN)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Site decided not to open this study
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Dr Stephen Chia, British Columbia Cancer Agency
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: OZM-003
Record Dates: First submitted 2008-02-14; First posted 2008-03-03 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2010-11

CONDITIONS: Locally Advanced Squamous Cell Carcinomas of the Head and Neck (SCCHN)
Keywords: squamous cell carcinoma; head and neck; Neoadjuvant Sorafenib and Concurrent Sorafenib, Cisplatin and Radiation
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Sorafenib; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment Group 1: Cohort 1 (Experimental): Cohort 1 - sorafenib 200 mg PO bid concurrent with radiation
  Interventions: Drug: sorafenib
- Treatment Group 1: sorafenib and radiation: Cohort 2 (Experimental): Cohort 2 - sorafenib 400 mg PO bid concurrent with radiation
  Interventions: Drug: sorafenib
- Treatment Group 2: Cohort 3 (Experimental): Cohort 3 - sorafenib 200 mg PO bid / cisplatin 75 mg/m2 weeks 1, 4 and 7
  Interventions: Drug: sorafenib and cisplatin
- Treatment Group 2: Cohort 4 (Experimental): o Cohort 4 - sorafenib 400 mg PO bid/ cisplatin 75 mg/m2 weeks 1, 4 and 7
  Interventions: Drug: sorafenib and cisplatin
- Treatment Group 2:Cohort 5 (Experimental): Cohort 5 - sorafenib 400 mg PO bid/ cisplatin 100 mg/m2 weeks 1, 4 and 7
  Interventions: Drug: sorafenib and cisplatin

INTERVENTIONS:
Drug: sorafenib — Cohort 1 - sorafenib 200 mg PO bid concurrent with radiation
  Arms: Treatment Group 1: Cohort 1
Drug: sorafenib — o Cohort 2 - sorafenib 400 mg PO bid concurrent with radiation
  Arms: Treatment Group 1: sorafenib and radiation: Cohort 2
Drug: sorafenib and cisplatin — Cohort 3 - sorafenib 200 mg PO bid / cisplatin 75 mg/m2 weeks 1, 4 and 7
  Arms: Treatment Group 2: Cohort 3
Drug: sorafenib and cisplatin — o Cohort 4 - sorafenib 400 mg PO bid/ cisplatin 75 mg/m2 weeks 1, 4 and 7
  Arms: Treatment Group 2: Cohort 4
Drug: sorafenib and cisplatin — Cohort 5 - sorafenib 400 mg PO bid/ cisplatin 100 mg/m2 weeks 1, 4 and 7
  Arms: Treatment Group 2:Cohort 5

SUMMARY:
The purpose of this study is to assess the safety and determine MTD (maximal tolerated doses) and recommended doses of neoadjuvant sorafenib (BAY 43-9006) and concurrent sorafenib, cisplatin and radiation in the locally advanced squamous cell carcinomas of the head and neck (SCCHN)patient population.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the head and neck is a relatively common malignancy in both Canada and the United States. Despite advancements made with the demonstration of improved outcomes for concurrent platinum based chemotherapy with radical radiation in locally advanced SCCHN, approximately 50% of cases will recur. The current treatment of locoregionally recurrent/metastatic SCCHN is palliative in intent, with a median survival in this population of 6-8 months. Thus improvements to the current backbone treatment of locally advanced SCCHN, that is platinum based chemotherapy with radical radiation, are desperately needed.

This is a non-randomized, open-label, phase I dose escalation trial of neoadjuvant Sorafenib and concurrent Sorafenib, Cisplatin and radiation in locally advanced squamous cell carcinomas of the head and neck (SCCHN).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: Treatment Group 1 (Cohorts 1 & 2) - Radiation and Sorafenib Only.

1. Previously untreated squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx. Histological or cytological confirmation is required. The disease must be considered to be potentially curable with radiation only.
2. Stage III or IV disease (UICC/AJCC classification, 6th edition)
3. Age ≥18
4. Patients for whom concurrent cisplatinum is contraindicated due to poor patient tolerance (significant weight loss > 10% of body weight, mild renal dysfunction, ototoxicity, neuropathy, or age >70) yet deemed fit for radical radiation.
5. Signed written consent.
6. Availability for follow-up after treatment.
7. If the patient is fertile he/she is aware of the risk of becoming pregnant or fathering children and will use adequate contraception (oral contraception, IUD, diaphragm and spermicide or male condom and spermicide) throughout therapy and for at least 2 weeks after therapy.
8. Life expectancy greater than 6 months

Inclusion Criteria: Treatment group 2 (Cohorts 3 to 5) - Radiation, Sorafenib and Cisplatin.

1. Previously untreated squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx. Histological or cytological confirmation is required. The disease must be considered to be potentially curable by combined chemoradiation.
2. Stage III or IV disease (UICC/AJCC classification, 6th edition)
3. Age ≥18.
4. Signed written consent.
5. Availability for follow-up after treatment.
6. If the patient is fertile, he/she is aware of the risk of becoming pregnant or fathering children and will use adequate contraception (oral contraception, IUD, diaphragm and spermicide or male condom and spermicide) throughout therapy and for at least 3 months after therapy.
7. Life expectancy greater than 6 months

Exclusion Criteria:

Treatment Group 1 (Cohorts 1 & 2) - Radiation and Sorafenib Only.

1. ECOG performance status 3 or 4
2. Absolute neutrophil count <1.0 X 109/L, platelet count <100 X 109/L or hemoglobin <90 g/L.
3. Serum bilirubin ≥1.5 times ULN or AST/ALT ≥ 2.5 times ULN.
4. Calculated creatinine clearance (Cockcroft-Gault) <40 mL/min. For patients in whom the calculated creatinine clearance is borderline, GFR may be estimated by nuclear renogram with the creatinine clearance ≥ 40 mL/min to be eligible.
5. Uncontrolled hypertension despite adequate anti-hypertensive medications
6. Bleeding diathesis
7. Significant inter-current illness that will interfere with the radiation therapy during the trial such as HIV infection, pulmonary compromise, active significant alcohol abuse, active infection or febrile illness
8. Any history of myocardial infarction, congestive heart failure (NY Heart Association Class 3 or 4), any history of ventricular arrhythmias, angina or active coronary heart disease within 6 months.
9. Primary cancers of the nasal and paranasal cavities, and of the nasopharynx.
10. Evidence of distant metastases. If based on the best available clinical evidence the investigator wishes to enroll the subject on trial, discussion and documentation with one of the principal investigators is required.
11. Weight loss greater than 25% of usual body weight in the 3 months preceding trial entry.
12. High risk for poor compliance with therapy or follow-up as assessed by investigator.
13. Pregnant or lactating women.
14. Prior radiation therapy to greater than 30% of the bone marrow
15. Prior experimental therapy for cancer within 30 days of entering the trial.
16. Prior radiation for head and neck cancer.
17. Patients with prior cancers, except: those diagnosed more than five years ago with no evidence of disease recurrence and a clinical expectation of recurrence of less than 5%; or successfully treated non-melanoma skin cancer; or carcinoma in situ of the cervix. However, any patient with previous invasive breast cancer, prostate cancer or melanoma is excluded.

Exclusion Criteria: Treatment group 2 (Cohorts 3 to 5) - Radiation, Sorafenib and Cisplatin.

1. ECOG performance status 3 or 4
2. Absolute neutrophil count <1.0 X 109/L, platelet count <100 X 109/L or hemoglobin <90 g/L.
3. Serum bilirubin ≥1.5 times ULN or AST/ALT ≥ 2.5 times ULN.
4. Calculated creatinine clearance (Cockcroft-Gault) <55 mL/min. For patients in whom the calculated creatinine clearance is borderline, GFR may be estimated by nuclear renogram with the creatinine clearance ≥ 55 mL/min to be eligible.
5. Uncontrolled hypertension despite adequate anti-hypertensive medications
6. Bleeding diathesis
7. Significant inter-current illness that will interfere with the chemotherapy or radiation therapy during the trial such as HIV infection, cardiac insufficiency, pulmonary compromise, active significant alcohol abuse, active infection or febrile illness,
8. Any history of myocardial infarction, any history of ventricular arrhythmias, angina or active coronary heart disease within 6 months. Significant cardiac disease resulting in an inability to tolerate the intravenous fluid load as required for administration of cisplatin.
9. Primary cancers of the nasal and paranasal cavities, and of the nasopharynx.
10. Evidence of distant metastases. If based on the best available clinical evidence the investigator wishes to enroll the subject on trial, discussion and documentation with one of the principal investigators is required.
11. Symptomatic peripheral neuropathy ≥ grade 2.
12. Clinically significant sensori-neural hearing impairment which may be exacerbated by cisplatin (audiometric abnormalities without corresponding clinical hearing impairment will not be grounds for exclusion)
13. Weight loss greater than 20% of usual body weight in the 3 months preceding trial entry.
14. High risk for poor compliance with therapy or follow-up as assessed by investigator.
15. Pregnant or lactating women.
16. Prior radiation therapy to greater than 30% of the bone marrow
17. Prior experimental therapy for cancer within 30 days of entering the trial.
18. Prior radiation for head and neck cancer.
19. Patients with prior cancers, except: those diagnosed more than five years ago with no evidence of disease recurrence and a clinical expectation of recurrence of less than 5%; or successfully treated non-melanoma skin cancer; or carcinoma in situ of the cervix. However, any patient with previous invasive breast cancer, prostate cancer or melanoma is excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To assess the safety of neoadjuvant BAY 43-9006 (sorafenib) and concurrent BAY 43-9006 with radiation in a cohort of SCCHN | ongoing

SECONDARY OUTCOMES:
MTD Maximal tolerated dose | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chia, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada